CLINICAL TRIAL: NCT02894307
Title: Evaluation of Thromboembolic Events in Patients With Bileaflet Mechanical Valves in Mitral Position Before and After Rivaroxaban Use: RMV Study
Brief Title: Rivaroxaban in Mechanical Valves: RMV Study
Acronym: RMV
Status: No longer available | Type: Expanded Access
Sponsor: Hospital Ana Nery (Other)
Collaborators: Federal University of Bahia (Other)
Responsible Party: Principal Investigator, Andre Duraes, MD, PhD, Prof Dr Andre Duraes, Hospital Ana Nery
Other Study IDs: 69327617.7.0000.5028
Record Dates: First submitted 2016-09-05; First posted 2016-09-09 (Estimated); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Prosthesis; Cardiac, Heart, Functional Disturbance as Result
Keywords: Mechanical prosthesis; Rivaroxaban
MeSH Terms: interventions — Rivaroxaban

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Rivaroxaban — In patients with mechanical valves and unstable INR
  Other Names: Xarelto 15 mg

SUMMARY:
Anticoagulant treatment reduces the incidence of death and cardioembolic events in patients with atrial ﬁbrillation or prosthetic heart valve and the incidence of death and recurrences in patients with VTE. Warfarin and similar vitamin K antagonists (VKA) have been the standard therapy for patients with a metallic valve, or bioprosthesis with atrial fibrillation (AF). The Dabigatran versus Warfarin in Patients with Mechanical Heart Valves (RE-ALIGN) trial comparing dabigatran etexilate to warfarin was the only randomized controlled study in patient with mechanical valve prosthesis, but it was terminated prematurely because of an excess of thromboembolic and bleeding events among patients in the dabigatran group. To date, novel oral anticoagulants (NOACs) have shown to be not both safe and or effective for patients with mechanical valves.

DETAILED DESCRIPTION:
Anticoagulant treatment reduces the incidence of death and cardioembolic events in patients with atrial ﬁbrillation or prosthetic heart valve and the incidence of death and recurrences in patients with VTE.

Warfarin and similar vitamin K antagonists (VKA) have been the standard therapy for patients with a metallic valve, or bioprosthesis with atrial fibrillation (AF). Warfarin works by binding to vitamin K epoxide reductase to inhibit vitamin K-dependent coagulation factors II, VII, IX, and X. For all its extensive use, warfarin has many clinical shortcomings, including variable pharmacokinetic and pharmacodynamics properties, a narrow therapeutic index range, and numerous interactions with certain foods and drugs. All of these factors contribute to the need for frequent coagulation laboratory monitoring and dosage adjustments.

Even with the appropriate use of therapy, the incidence of thromboembolic events is still substantial: 1-4% per year. Furthermore, bleeding risk is significant, ranging from 2% to 9% per year. The VKA's narrow therapeutic index and they have a complex pharmacology, e.g. long pharmacologic inertia and the common interaction with other drugs. These features make the management of these drugs a challenge for physicians and their patients.

The Dabigatran versus Warfarin in Patients with Mechanical Heart Valves (RE-ALIGN) trial comparing dabigatran etexilate to warfarin was the only randomized controlled study in patient with mechanical valve prosthesis, but it was terminated prematurely because of an excess of thromboembolic and bleeding events among patients in the dabigatran group. Most thromboembolic events among patients in the dabigatran group occurred in population A (patients who had started a study drug within 7 days after valve surgery), with fewer occurring in population B (patients who had undergone valve implantation more than 3 months before randomization). Besides, stroke, death and major bleeding occurred only in population A. In this study, rivaroxaban will be used in patients with mechanical valves and unstable INR in a before and after designed.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 64 years at entry;
* Patients with mitral mechanical valve for at least 3 months postoperatively;
* Brain computed tomography scan without hemorrhage or findings of acute cerebral infarction on the last 2 days of screening;
* Exclusion of atrial thrombus or valve prosthesis thrombosis by transesophageal echocardiograph on the last 2 days of screening;
* Written, informed consent;

Exclusion Criteria:

* Previous hemorrhagic stroke;
* Ischemic stroke in the last 6 months;
* Renal impairment (creatinine clearance rates < 50 ml/min);
* Active liver disease (any etiology);
* Concomitant use of any antiplatelet (aspirin, clopidogrel, prasugrel, ticagrelor, ticlopidine, etc);
* Increased risk of bleeding (congenital or acquired);
* Uncontrolled hypertension;
* Gastrointestinal hemorrhage within the past year;
* Anemia (hemoglobin level <10 g/dL) or thrombocytopenia (platelet count < 100 × 109/L);
* Active infective endocarditis;
* Pregnant or lactating women;

Ages: 18 Years to 64 Years | Sex: All
Age Groups: Adult

REFERENCES:
- [Result] Duraes AR, de Souza Roriz P, de Almeida Nunes B, Albuquerque FP, de Bulhoes FV, de Souza Fernandes AM, Aras R. Dabigatran Versus Warfarin After Bioprosthesis Valve Replacement for the Management of Atrial Fibrillation Postoperatively: DAWA Pilot Study. Drugs R D. 2016 Jun;16(2):149-54. doi: 10.1007/s40268-016-0124-1. PMID 26892845
- [Derived] Duraes AR, Bitar YSL, Lima MLG, Santos CC, Schonhofen IS, Filho JAL, Roever L. Usefulness and Safety of Rivaroxaban in Patients Following Isolated Mitral Valve Replacement With a Mechanical Prosthesis. Am J Cardiol. 2018 Sep 15;122(6):1047-1050. doi: 10.1016/j.amjcard.2018.06.015. Epub 2018 Aug 8. PMID 30098707